CLINICAL TRIAL: NCT02180100
Title: A Randomized, Parallel-group Study of Terconazole Vaginal Suppository vs Fluconazole for the Treatment of Severe
Brief Title: Terconazole Vaginal Suppository vs Fluconazole for the Treatment of Severe Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Collaborators: Shanghai Shyndec Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shangrong Fan, Prof of Obstetrics and Gynecology, Peking University Shenzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUSH-GNY-2013-01
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Terconazole Vaginal Suppository (Experimental): Terconazole Vaginal Suppository inserted intravaginally once daily before bedtime for 6 consecutive days
  Interventions: Drug: Terconazole Vaginal Suppository
- Fluconazole (Active Comparator): orally Fluconazole 150 mg (Pfizer Pharmaceuticals) at day 1 and day 4.
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Terconazole Vaginal Suppository — Terconazole Vaginal Suppository inserted intravaginally once daily before bedtime for 6 consecutive days
  Other Names: Tekangzuo Yindao Shuan
  Arms: Terconazole Vaginal Suppository
Drug: Fluconazole — orally Fluconazole 150 mg (Pfizer Pharmaceuticals) at day 1 and day 4.
  Other Names: Diflucan
  Arms: Fluconazole

SUMMARY:
The objectives of this study were to demonstrate comparable safety and efficacy of Terconazole Vaginal Suppositories, 80 mg and fluconazole in the treatment of subjects with severe vulvovaginal candidiasis.

DETAILED DESCRIPTION:
This study were to demonstrate comparable safety and efficacy of Terconazole Vaginal Suppository 80 mg inserted intravaginally once daily before bedtime for 6 consecutive days and oral fluconazole 150mg at day 1 and day 4 in the treatment of subjects with severe vulvovaginal candidiasis.

ELIGIBILITY:
Inclusion Criteria:

* Vulvovaginal candidiasis infection is diagnosed, the symptoms evaluated using a numerical rating system based on severity (absent=0; mild=1; moderate=2; severe=3) with a minimum VVC Composite Signs/Symptoms score of 7
* Subject completes the informed consent process
* Subject agrees to take study medication when scheduled
* Subject complies with all clinical trial instructions. Commits to all follow-up visits
* Subject agrees to abstain from sexual intercourse from the time of randomization through the first seven days immediately following treatment

Exclusion Criteria:

* had any other sexually transmitted disease or gynaecological abnormality requiring treatment
* had a disease known to predispose to candidiasis such as diabetes mellitus, or were receiving antibiotics or corticosteriods
* had used antifungal medication in the week before entry; or
* were expected to menstruate within seven days of the start of treatment
* infected more than one candida species

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shangrong Fan, M.D., Principal Investigator — Peking University Shenzhen Hospital
Locations (1):
- Peking University Shenzhen Hosptal, Shenzhen, Guangdong, China

REFERENCES:
- [Result] Li T, Zhu Y, Fan S, Liu X, Xu H, Liang Y. A randomized clinical trial of the efficacy and safety of terconazole vaginal suppository versus oral fluconazole for treating severe vulvovaginal candidiasis. Med Mycol. 2015 Jun;53(5):455-61. doi: 10.1093/mmy/myv017. Epub 2015 Apr 15. PMID 25877666
- See also: Terconazole Vaginal Suppository vs Fluconazole for the Treatment of Severe Vulvovaginal Candidiasis — http://www.ncbi.nlm.nih.gov/pubmed/25877666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At Clinic
Period: Overall Study
Arm/Group | Terconazole Vaginal Suppository | Fluconazole
Started | 70 | 70
Completed | 58 | 66
Not Completed | 12 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Terconazole Vaginal Suppository | Fluconazole | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 70 | 140
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 70 | 140
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mycological Cure 1
Description: Based on candida culture
Time Frame: Between day 7-14 after treatment, an average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Terconazole Vaginal Suppository | Fluconazole
Number analyzed (Participants) | 58 | 66
Participants | 46 | 47

2. Secondary Outcome: Mycological Cure 2
Description: Based on Candida culture
Time Frame: Between day 28-35 after treatment, an average of 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Terconazole Vaginal Suppository | Fluconazole
Number analyzed (Participants) | 58 | 66
Participants | 36 | 35

ADVERSE EVENTS:
Time Frame: Day 35 after treatment
Description: Vulvovaginal pruritus, burning and irritation
Arm/Group | Terconazole Vaginal Suppository | Fluconazole
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less